CLINICAL TRIAL: NCT03143543
Title: Phase I Functional Magnetic Resonance Imaging (fMRI) Pharmacodynamic Studies of Compounds for Opioid Use Disorder and Cocaine Use Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA removal of drug from the market due to cancer risks
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20003329; 5U54DA038999-04 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2017-05-08 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2019-07

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders
Keywords: cocaine disorder; opioid disorder; lorcaserin; MRI; fMRI
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Intervention Model Description: Starting lorcaserin dosage of 10 mg per day for 7 days in one arm, versus placebo for 7 days in parallel arm. An interim analysis will take place after 15 subjects have completed at each arm. Based on the interim analysis, if there is no significant effect and no trend towards significance for the lower dose of lorcaserin in the primary regions of interest for fMRI task, and no significant accumulation of adverse effects, testing will stop for the lower dose of lorcaserin, and testing will begin for the higher dose, which is the FDA approved usual dose for lorcaserin (20 mg per day, given as 10 mg twice per day). The higher dose of lorcaserin will be tested in a two group parallel arm design, initially with 15 subjects in lorcaserin arm and 15 subjects in the parallel placebo arm. Another interim analysis will take place after 15 subjects have completed at each arm in the higher dose lorcaserin study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A Lorcaserin (10mg) (Experimental): 10 mg lorcaserin orally for 7 days
  Interventions: Drug: Group A Lorcaserin (10mg)
- Group B Parallel Placebo (Placebo Comparator): Placebo orally for 7 days vs Group A
  Interventions: Other: Group B Parallel Placebo
- Group A2 Lorcaserin (20 mg) (Experimental): 20 mg lorcaserin orally for 7 days
  Interventions: Drug: Group A2 Lorcaserin (20 mg)
- Group B2Parallel Placebo (Placebo Comparator): Placebo orally for 7 days vs Group A2
  Interventions: Other: Group B2 Parallel Placebo

INTERVENTIONS:
Drug: Group A Lorcaserin (10mg) — 10 mg lorcaserin orally for 7 days
  Other Names: Belviq
  Arms: Group A Lorcaserin (10mg)
Drug: Group A2 Lorcaserin (20 mg) — 20 mg lorcaserin orally for 7 days
  Other Names: Belviq
  Arms: Group A2 Lorcaserin (20 mg)
Other: Group B Parallel Placebo — Oral placebo vs 10 mg lorcaserin
  Arms: Group B Parallel Placebo
Other: Group B2 Parallel Placebo — Oral placebo vs 20 mg lorcaserin
  Arms: Group B2Parallel Placebo

SUMMARY:
The purpose of Project 2 is to execute phase I functional magnetic resonance imaging (fMRI) studies to assess the effects of lorcaserin on brain target engagement (measured by fMRI brain activation and neural connectivity) in cocaine use disorder (CocUD) subjects and/or opioid use disorder.

DETAILED DESCRIPTION:
During the screening period (Study Days -3 and -2), the urine drug screen (UDS) must be negative for cocaine and opioids, and the self-reported last use of cocaine or opioids must be at least seven days prior to this result, in order to ensure that possible cocaine or opioid withdrawal has ended. After these criteria have been met, all subjects will receive placebo at 8:30 AM for one day during the Placebo Pretreatment Baseline Day (Study Day -1). The first fMRI session (fMRI #1) will take place at 10:00 AM on the following day (Study Day 1). Following fMRI #1, the subjects will be randomized into two parallel groups (Group A: Lorcaserin; Group B: Parallel Placebo). Based on the information that a lower dose of lorcaserin has the potential to be clinically effective , and based on the safety and abuse potential data from human studies, as well as the preclinical data on interaction with cocaine , the study will begin with the lower dose of lorcaserin (10 mg per day). For Group A (lorcaserin group), the lorcaserin dose will be 10 mg orally per day for 7 days. For Group B (parallel placebo group), identical appearing placebo will be given orally according to the same schedule as lorcaserin for 7 days. After the 7 days of treatment with study medications, fMRI #2 will take place, then study medications will be discontinued. A follow-up visit will occur one week after the last dose of study medication. See Section II.b for details and criteria for stopping or continuing this dosage based on the results of the interim analysis, which will take place after 15 subjects have completed at each arm. Based on the interim analysis, if there is no significant effect and no trend towards significant effect (p > 0.10) for the lower dose lorcaserin in the primary regions of interest for the cue-reactivity fMRI task, and no significant accumulation of adverse effects, then testing will stop for the lower dose of lorcaserin, and testing will begin for the higher dose of lorcaserin (10 mg twice per day) 7 days. The higher dose of lorcaserin will be tested in a two group parallel arm design, initially with 15 subjects in the high dose lorcaserin arm and 15 subjects in the parallel placebo arm. Another interim analysis will take place after 15 subjects have completed at each arm in the higher dose lorcaserin study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females treatment-seeking cocaine and/or opioid users between 18 and 55 years of age
2. Understand the study procedures and provide written informed consent
3. Must be in residential treatment for substance use disorder
4. Meet current DSM-5 criteria for Cocaine Use Disorder with moderate or severe severity, and current DSM-IV diagnosis of Cocaine Dependence or Abuse, and/or current DSM-5 criteria for Opioid Use Disorder with moderate or severe severity, and/or current DSM-IV diagnosis of Opioid Dpendence or Abuse.
5. Have been abstinent from cocaine and/or opioid use for at least 1 week
6. Have vital signs as follows: resting pulse between 55 and 95 bpm, blood pressures between 90-139 mm Hg systolic and 50-89 mm Hg diastolic
7. Have hematology and chemistry laboratory tests that are within normal limits, except that liver function tests must be less than twice the upper limit of normal and judged by the study physician to be clinically insignificant.
8. Have a normal baseline ECG as shown by normal sinus rhythm with the exception of sinus arrhythmia or mild sinus bradycardia (heart rate 50-59 beats per minute), and with normal conduction (including normal QTcF) with the exception of early repolarization judged to be clinically insignificant by both the study physician and the study cardiologist.
9. For adults who ar 20 years old or older, have a Body Mass Index (BMI) that is 18.5 or greater according to the CDC Calculator for Adults.. For adolescents who are 18 or 19 years old, BMI that is fifth percentile or greater according to the CDC Calculator for Children and Teens.
10. Have no contraindications for study participation as determined by history and physical examination
11. Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory and fMRI testing
12. No pregnant or nursing women will be permitted in the study, and women must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device with spermicide, or condoms). Men will be advised to use condoms. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and at the end of study participation.

Exclusion Criteria:

1. Have concurrent DSM-IV diagnosis of any psychoactive substance use dependence other than cocaine, nicotine, marijuana, or opioid dependence.
2. Have a DSM-5 axis I psychiatric disorder, other than substance use disorder, including by not limited to Bipolar Disorder, Major Depressive Disorder, ADHD, or Schizophrenia, or a neurological disorder requiring ongoing treatment and/or making study participation unsafe.
3. Subjects with evidence or history of any clinically significant medical disorder including cardiovascular, pulmonary, CNS, hepatic, or renal, except that controlled hypertension, controlled hypothyroidism, and cancer in remission will not be excluded.
4. Subjects who have Type 1 or Type 2 diabetes mellitus, since weight loss may increase the risk of hypoglycemia in patients with Type 2 diabetes mellitus treated with insulin secretagogues (eg., sulfonylureas), and lorcaserin has not been studied in combination with insulin.
5. Subjects with an abnormal QTcF on ECG
6. Have a history of seizures (excluding childhood febrile seizures), or loss of consciousness for more than 20 minutes
7. Have significant current suicidal or homicidal ideation or a suicide attempt within the past 6 months
8. Be HIV positive by self-report or history
9. Be pregnant or nursing or not using a reliable form of contraception if able to conceive. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and at the end of study participation
10. Have an other illness or condition, which in the opinion of the PI would preclude safe and/or successful completion of the study.
11. Be using any medications or drugs that can affect the central nervous system other than cocaine, marijuana, alcohol, caffeine, and nicotine.
12. Be using any medication (including over-the-counter medication or food suplements) that may interact adversely with lorcaserin, including other serotonergic drugs, including SNRIs and SSRIs, triptans, drugs that impair metabolism of serotonin (including MAOIs), dietary supplements such as St. John's wort and tryptophan, tramadol, or antipsychotics or other dopamine antagonists.. See Lorcaserin Drug Interactions table (attached) for detailed list of these medications.
13. Prior to starting study medication, and prior to each MRI scanning session, have positive breath alcohol level, or have a positive urine drug screen for any drug of abuse other than marijuana.
14. Have metal fragments or other bodily metal (e.g., pacemaker), or significant claustrophobia that would put the subjects at risk for MRI scanning.
15. Subjects who are allergic to lorcaserin
16. Subjects who have taken any investigational drug within 90 days prior to baseline.
17. Subjects who are taking opioids for medical reasons (e.g., cancer, injuries, etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Target engagement by lorcaserin | Seven Days
  To determine target engagement by lorcaserin in a cocaine-Stroop and/or opioid-Stroop cue-reactivity fMRI task in cocaine use disorder (CocUD) and/or Opioid Use Disorder Subjects

CONTACTS AND LOCATIONS:
Overall Officials: James Bjork, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No